CLINICAL TRIAL: NCT02903485
Title: Bypassing Anesthesiologist Assessment Before Cataract Surgery: a Non Inferiority Study
Acronym: CATARIDE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: JMD_2014-31
Record Dates: First submitted 2016-09-08; First posted 2016-09-16 (Estimated); Last update posted 2018-12-07 (Actual); Status verified 2017-11

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- nurses (intervention arm) (Experimental): for patients without risk factors, the anesthetic team is not involved in patients' care
  Interventions: Other: nurses perform presurgical assessement and surveillance during surgery
- anesthetic team (control arm) (Active Comparator): the anesthetic team is involved in every patient's care (with or without risk factors)
  Interventions: Other: the anesthetic team performs presurgical assessement and surveillance during surgery

INTERVENTIONS:
Other: nurses perform presurgical assessement and surveillance during surgery
  Arms: nurses (intervention arm)
Other: the anesthetic team performs presurgical assessement and surveillance during surgery
  Arms: anesthetic team (control arm)

SUMMARY:
This study aims to demonstrate that presurgical assessement of patients' risk factors and surveillance during surgery, both performed by nurses, are not inferior to anesthetic team's care, concerning the rate of complications in cataract surgery with topical anesthesia.

The nurse performs the triage of patients based on a chart of risk factors assessment. The triage, according to the presence or not of risk factors, leads to patients' care by an anesthetic team (medical anesthesist for pre-surgical assessement and anesthetic nurse for surveillance during surgery) or to patients' pre-surgical assessement and surveillance during surgery both performed only by nurses.

In the control group, all patients are taken care of by an aesthetic team, with medical pre surgical assessement and surveillance during surgery both performed by anesthetic nurses.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years old
* cataract surgery scheduled with topical anesthetics
* outpatient surgery

Exclusion Criteria:

* presurgical nurse assessment leading to the need for the anesthetic staff presence during surgery
* general, peribulbar or other locoregional anesthesia required by patient's condition
* concomitant surgery planified (glaucoma, vitrectomy…)
* patient's refusal to participate in the study
* no health insurance coverage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 578 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Incidence of complications | through study completion, up to 6 months
  complications occuring in operating theatre include systolic blood pressure > 200 mmHg or < 80 mmHg, diastolic blood pressure > 110 mmHg, heart rate < 45/mn for at least 1 mn, oxygen saturation (SpO2) <90% for at least 1 mn, impossibility to start or to pursue surgery because of patient condition.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel Devys, MD, Principal Investigator — Fondation Ophtalmologique Adolphe de Rothschild
Locations (1):
- Fondation Ophtalmologique Adophe de Rothschild, Paris, France